CLINICAL TRIAL: NCT05229042
Title: An Exploratory Study to Investigate the Safety and Efficacy of Ricolinostat for Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Brief Title: A Study to Investigate the Safety and Efficacy of Ricolinostat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing 3E-Regenacy Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCRG-CN-101
Record Dates: First submitted 2022-01-19; First posted 2022-02-08 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Nervous System Diseases
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — ricolinostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blank
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active arm (Active Comparator): Subjects received ricolinostat
  Interventions: Drug: Ricolinostat
- Placebo arm (Placebo Comparator): Subjects received placebo
  Interventions: Drug: Ricolinostat

INTERVENTIONS:
Drug: Ricolinostat — Oral
  Other Names: Placebo

SUMMARY:
This is a double-blind, placebo-controlled study during which patients will receive ricolinostat or placebo.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled study during which patients will receive ricolinostat or placebo.

Prior to randomization, patients will participate in the Screening and Baseline assessment period to ensure that they meet study inclusion/exclusion criteria.

Following the Screening and Baseline assessment period, patients who meet entry criteria will be randomized in a 2:1 ratio to receive either ricolinostat or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study's purpose and requirements, and able to voluntarily provide informed consent to participate.
2. Age ≥ 18 years and < 70 years at the time of signing the informed consent form (ICF).
3. Female patients diagnosed with breast cancer:

   1. Who have been treated with either docetaxel or paclitaxel.
   2. Who have a Karnofsky performance status of 70 or more at Screening.
   3. Who have completed their chemotherapy at least 1 month prior to randomization.
4. Neuropathy of <Grade 4 using the general guideline of grading scales defined in Common Terminology Criteria for Adverse Events (CTCAE; v5.0) .
5. Women of childbearing potential (WOCBP) must agree to use reliable contraceptive methods for the duration of the study and for at least 3 months after completing treatment with study drug. For the purposes of this study, reliable methods of contraception include abstinence, oral contraceptives, hormonal contraceptive implants such as Nexplanon, hormonal vaginal ring such as NuvaRing, intrauterine devices in place for at least 3 months, or barrier methods used in conjunction with spermicide. To be considered post-menopausal and of non childbearing potential, women less than 60 years with less than 2 years since their last period must have follicle-stimulating hormone (FSH) > 40 IU/L and estradiol < 20 pg/mL unless on hormone replacement.
6. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Women who are pregnant or lactating.
2. Extremely overweight, defined as body mass index (BMI) > 40 kg/m2.
3. Presence of any neuropathy other than CIPN.
4. Presence of a clinical condition commonly associated with neuropathy that could better account for the presence of the patient's neuropathy, such as diabetes or a risk factor for marked B12 deficiency (malabsorption syndrome, atrophic gastritis, strict vegan diet, etc.), or a megaloblastic (macrocytic) anemia consistent with B12 deficiency.
5. Presence of skin conditions in the affected dermatome that, in the judgement of the Investigator, could interfere with evaluation of the neuropathic pain condition.
6. Presence of non-CIPN pain that may interfere with study assessments and/or self-evaluation of peripheral neuropathic pain.
7. History of alcoholism or drug/chemical abuse within 1 year prior to randomization as judged by the Investigator based on clinical history.
8. Opioid use at a dose of ≥ 30 morphine milligram equivalents on 3 or more days a week during the month at Screening.
9. The use of cannabidiol (CBD) during the 1 month at Screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
TEAT | 6 months
  The primary endpoint is the incidence of treatment-emergent adverse events (TEAEs) during the Treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Binhe Xue, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Beijing3ERegenacy, Beijing, China

IPD SHARING:
Plan to Share IPD: No